CLINICAL TRIAL: NCT01010464
Title: Effect of an Adhesion Reduction Plan on Enteric Adhesions, Obstruction, and Fistulae in the Management of the Surgical Open Abdomen: A Prospective, Randomized Clinical Trial in Trauma and Emergency General Surgery
Brief Title: An Adhesion Reduction Plan in the Management of the Surgical Open Abdomen
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Principal Investigator, William Chiu, Associate Professor of Surgery, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HP-00043289
Record Dates: First submitted 2009-11-09; First posted 2009-11-10 (Estimated); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Open Abdomen
Keywords: Adhesions; Open abdomen; Laparotomy
MeSH Terms: conditions — Tissue Adhesions | interventions — Seprafilm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adhesion Reduction Plan (Experimental): Lysis of adhesions and application of Seprafilm
  Interventions: Procedure: Adhesion Reduction Plan
- Standard Management (No Intervention): Standard management and no application of Seprafilm

INTERVENTIONS:
Procedure: Adhesion Reduction Plan — Lysis of adhesions and application of a minimum of 4 sheets of a sodium hyaluronate-based bioresorbable membrane
  Other Names: Seprafilm
  Arms: Adhesion Reduction Plan

SUMMARY:
The purpose of this study is to determine whether an adhesion reduction plan, consisting of early adhesion prevention and application of a bioresorbable membrane is effective in reducing the severity of adhesions and the incidence of complications in managing the open abdomen in trauma and emergency general surgery.

DETAILED DESCRIPTION:
Adhesions are a common consequence of abdominal surgery. Trauma and emergency general surgery patients may require an open abdomen and undergo a series of abdominal operations, which may be increasingly complicated by the presence of adhesions. Adhesions appear soon after the initial operation and gradually mature within days. The effects of adhesion development on subsequent surgery may include: increased procedure time; difficulty differentiating, exposing, and accessing tissue planes; and increased risk of inadvertent enterotomy. Complications of adhesions include enteric obstruction and enterocutaneous fistulae. This study will determine whether an adhesion reduction plan, consisting of early adhesion prevention and application of a bioresorbable membrane is effective in reducing the extent and severity of adhesions and the incidence of complications in managing the open abdomen in trauma and emergency general surgery.

ELIGIBILITY:
Inclusion Criteria:

* Trauma patients with open abdomen after initial laparotomy
* Emergency surgery patients with open abdomen after initial laparotomy
* Able to obtain consent from patient or LAR before any research initiated

Exclusion Criteria:

* Seprafilm application at initial laparotomy
* Patient is a prisoner
* Inability to obtain informed consent
* Consentable person does not speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-01; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Extent and severity of adhesions | Each abdominal re-entry and re-exploration

SECONDARY OUTCOMES:
Time for lysis of adhesions | Each abdominal re-entry and re-exploration
Incidence of complications | Hospital admission

CONTACTS AND LOCATIONS:
Overall Officials: William C. Chiu, M.D., Principal Investigator — University of Maryland, College Park
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States